CLINICAL TRIAL: NCT02282566
Title: A Pilot Trial to Assess the Effect of a Protein-Nutrition Beverage on Skeletal Muscle Protein Synthesis in Women
Brief Title: Effect of Protein-nutrition Beverages on Muscle Protein Synthesis in Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: PEP-1331
Record Dates: First submitted 2014-10-30; First posted 2014-11-04 (Estimated); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Muscle Protein Synthesis
Keywords: Muscle protein synthesis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Protein-nutrition beverage - Placebo (Placebo Comparator): : 8 oz protein-nutrition beverage 1
  Interventions: Other: Protein-nutrition beverage
- Protein-nutrition beverage - Beverage 2 (Experimental): 8 oz protein-nutrition beverage 2
  Interventions: Other: Protein-nutrition beverage
- Protein-nutrition beverage - Beverage 3 (Experimental): 8 oz protein-nutrition beverage 3
  Interventions: Other: Protein-nutrition beverage
- Protein-nutrition beverage - Beverage 4 (Experimental): 8 oz protein-nutrition beverage 4
  Interventions: Other: Protein-nutrition beverage

INTERVENTIONS:
Other: Protein-nutrition beverage — Intervention involves consumption of one protein-nutrition beverage after exercise bout and 2 times per day for 5 days thereafter

SUMMARY:
This study investigates whether a protein-nutrition beverage can increase muscle protein synthesis to a similar magnitude as a control beverage.

DETAILED DESCRIPTION:
Potential participants will be screened, and if eligible, invited to participate. Body composition and physical activity level will be assessed during the initiation visit. During the trial visits, women receive a protein-nutrition beverage; muscle protein synthesis is assessed via blood analytes and muscle biopsies at rest and after exercise. Statistical analysis includes mixed model regression approach with change in muscle protein synthesis as the primary outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Older women, 65 to 75 years of age
2. At least 5 years post-menopausal
3. Body mass index (BMI) 20.00-29.99 kg/m2
4. Maintenance of habitual diet, physical activity patterns, and body weight throughout the trial
5. Low to moderate habitual physical activity ( > 3500 but < 10,000 steps/d, no structured activity)
6. In general good health (stage I hypertension allowed - 140/90) on the basis of medical history; and taking no medication other than anti-hypertensives, selective serotonin-reuptake inhibitors, and/or statins (excluding simvastatin [Zocor] and atorvastatin [Lipitor])
7. Participant understands the study procedures and signs forms providing informed consent to participate in the study and authorization for release of relevant protected health information to the study investigator.
8. Participant can consume a protein drink in the allotted time frame of 10 minutes

Exclusion Criteria:

1. History or presence of clinically important renal or gastrointestinal disorders, diabetes mellitus (glucose >126 mg/dL, fingerstick) or metabolic disease, unstable arrhythmia, angina, taking anti-diabetic, anti-inflammatory, platelet inhibitor, or anti-coagulant medications.
2. Vegan
3. Smoker
4. Overt osteoporosis and/or osteopenia and/or sarcopenia as determined by DXA
5. High physical activity or participating in regular structured exercise (> 10,000 steps/d)
6. History of allergy, sensitivity, or strong dislike towards any of the components of the study products (dairy protein)
7. Use of an investigational drug product within the last 30 days
8. Having participated in an another infusion protocol in the past year
9. Individual has a condition the PI believes would interfere with her ability to provide informed consent, comply with the study protocol, or which might confound the interpretation of the study results or put the person at undue risk
10. Subject does not understand English

Ages: 65 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-01-06 (Actual); Primary Completion 2017-03-30 (Actual); Study Completion 2017-03-30 (Actual)

PRIMARY OUTCOMES:
Change (timei -baseline) of muscle protein synthesis at rest and following exercise in response to the protein-nutrition beverages compared to a control beverage | 0-3 hours post consumption and 5 days post consumptions

SECONDARY OUTCOMES:
Change (timei -baseline) of blood sample analytes at rest and following exercise in response to the protein-nutrition beverages compared to a control beverage | 0-3 hours post consumption and 5 days post consumptions

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Philips, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Devries MC, McGlory C, Bolster DR, Kamil A, Rahn M, Harkness L, Baker SK, Phillips SM. Leucine, Not Total Protein, Content of a Supplement Is the Primary Determinant of Muscle Protein Anabolic Responses in Healthy Older Women. J Nutr. 2018 Jul 1;148(7):1088-1095. doi: 10.1093/jn/nxy091. PMID 29901760
- [Derived] Devries MC, McGlory C, Bolster DR, Kamil A, Rahn M, Harkness L, Baker SK, Phillips SM. Protein leucine content is a determinant of shorter- and longer-term muscle protein synthetic responses at rest and following resistance exercise in healthy older women: a randomized, controlled trial. Am J Clin Nutr. 2018 Feb 1;107(2):217-226. doi: 10.1093/ajcn/nqx028. PMID 29529146